CLINICAL TRIAL: NCT02006888
Title: The Efficacy and Safety of IBI-10090 for the Treatment of Inflammation Associated With Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ICON Bioscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C13-04
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Inflammation; Cataracts
Keywords: Inflammation; cataract surgery
MeSH Terms: conditions — Inflammation; Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- IBI-10090 low dose (Experimental): IBI-10090 low dose
  Interventions: Drug: IBI-10090
- IBI-10090 med dose (Experimental): IBI-10090 med dose
  Interventions: Drug: IBI-10090
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBI-10090
  Other Names: Dexycu
  Arms: IBI-10090 low dose; IBI-10090 med dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether IBI-10090 injection is effective in the treatment of inflammation associated with cataract surgery.

DETAILED DESCRIPTION:
A double blinded randomized trial to assess the efficacy and safety of IBI-10090, in two separate doses as compared to placebo (ATEC carrier only sans dexamethasone)

ELIGIBILITY:
Inclusion Criteria:

1. The patient must provide written informed consent by signing the Informed Consent approved by the Institutional Review Board (IRB).
2. Male or female patients at least 40 years of age scheduled for unilateral cataract surgery by phacoemulsification with posterior chamber intraocular lens implantation.
3. The patient must demonstrate best corrected visual acuity (BCVA) of 20/30-20/200 (with glare testing, if necessary) in the study eye and better than 20/200 in the fellow eye.
4. The patient must be considered by the Investigator to have visual acuity potential greater than 20/30 in the study eye.
5. The patient must have a corneal endothelial cell count by specular microscopy in the study eye of at least 2000 cells/mm2 with normal cell morphology.
6. A female patient of childbearing potential (premenopausal by medical history) must have a negative pregnancy test on Day 0 and be using an effective method of birth control (although no birth control method is 100% effective, the following are considered effective means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception using either a condom or diaphragm with spermicidal gel, an intrauterine device, or contraceptive hormone implant or patch) from Screening for the duration of the study.
7. The patient must be willing and able to understand and comply with the study procedures and to communicate meaningfully with study personnel.

Key Exclusion Criteria:

1. Patients who have used any ocular, topical or oral corticosteroids within 7 days prior to Day 0.
2. Patients who have received a periocular corticosteroid injection in the study eye in the 3 months prior to screening.
3. Patients who have received any intravitreal corticosteroid delivery vehicle (e.g., Retisert, Ozurdex, Iluvien) in the study eye at any time.
4. Patients who anticipate requiring treatment with any corticosteroids by any route, except inhalation, during the study.
5. Patients with an allergy or hypersensitivity to dexamethasone.
6. Patients who are known steroid responders (corticosteroid-related intraocular pressure elevation in either eye).
7. Patients who have used topical ocular NSAIDs in the study eye within 15 days prior to Day 0.
8. Patients who have undergone prior intraocular (non-laser) surgery in the study eye within 6 months prior to screening.
9. Patients who have undergone prior intraocular laser surgery in the study eye within 3 months prior to screening.
10. Patients with planned intraocular or laser surgery in the study eye for the duration of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: howard franklin, md, Study Director — ICON Bioscience Inc
Locations (1):
- Hull Eye Center, Lancaster, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled into the study on 19 December 2013 and the last patient completed the study on 03 October 2014.
Groups:
- IBI-10090 Low Dose: IBI-10090 low dose
  IBI-10090
- IBI-10090 Med Dose: IBI-10090 med dose
  IBI-10090
Period: Overall Study
Arm/Group | IBI-10090 Low Dose | IBI-10090 Med Dose | Placebo
Started | 158 | 156 | 80
Completed | 122 | 122 | 58
Not Completed | 36 | 34 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBI-10090 Low Dose | IBI-10090 Med Dose | Placebo | Total
Number analyzed (Participants) | 158 | 156 | 80 | 394
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 17 | 99
  >=65 years | 117 | 115 | 63 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 70 (9) | 71 (9) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 69 | 39 | 183
  Male | 83 | 87 | 41 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 14 | 56
  Not Hispanic or Latino | 139 | 133 | 66 | 338
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 17 | 21 | 11 | 49
  White | 129 | 123 | 67 | 319
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 1 | 13
Region of Enrollment [Number; unit: participants]
  United States | 158 | 156 | 80 | 394

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anterior Chamber Cell Clearing
Description: The primary efficacy outcome is anterior chamber cell clearing in the study eye at Day 8. The slit lamp examination for anterior chamber cells (ACC) is a recognized way to measure inflammation in the anterior chamber. During the slit lamp examination, the number of anterior chamber cells are quantified and graded: grade 0 (absent, 0 cells), grade 1 (1 to 5 cells), grade 2 (6 to 15 cells), grade 3 (16 to 30+ cells), or grade 4 (hypopyon). Anterior chamber cell clearing occurs when all the ACC are absent (grade 0).
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | IBI-10090 Low Dose | IBI-10090 Med Dose | Placebo
Number analyzed (Participants) | 158 | 156 | 80
Participants | 99 | 103 | 20

ADVERSE EVENTS:
Arm/Group | IBI-10090 Low Dose | IBI-10090 Med Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/156 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/158 | 0/156 | 0/80
Other Adverse Events (participants affected / at risk) | 16/158 | 4/156 | 7/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI-10090 Low Dose (N=158) | IBI-10090 Med Dose (N=156) | Placebo (N=80)
Corneal decompensation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI-10090 Low Dose (N=158) | IBI-10090 Med Dose (N=156) | Placebo (N=80)
eye pain (Eye disorders) | 16 (16) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes